CLINICAL TRIAL: NCT01826045
Title: A Multi-center, Randomized, Double Blind, Placebo Control, Parallel Design, Phase 2a Trial to Evaluate the Efficacy and Safety of PGA (Poly-gamma Glutamic Acid) for the Fertile Women With Cervical Intraepithelial Neoplasia 1 (CIN1)
Brief Title: Efficacy and Safety Study of PGA (Poly-gamma Glutamic Acid) for Cervical Intraepithelial Neoplasia
Acronym: PGA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioLeaders Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMT2012-BL-PGA-01; 12335 (Other: Korea Food and Drug Administration)
Record Dates: First submitted 2013-03-29; First posted 2013-04-08 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Treatment of Cervical Intraepithelial Neoplasia(CIN1)
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — poly(gamma-glutamic acid)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Poly-gamma Glutamic Acid (Experimental): Patients with cervical intraepithelial neoplasia 1(CIN1) will be administered Poly-gamma Glutamic Acid for 4 weeks.
  Interventions: Drug: Poly-gamma Glutamic Acid
- Placebo (Placebo Comparator): Patients with cervical intraepithelial neoplasia 1(CIN1) will be administered placebo for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Poly-gamma Glutamic Acid
  Arms: Poly-gamma Glutamic Acid
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and the safety of PGA(Poly-gamma Glutamic Acid) for the the fertile women with Cervical Intraepithelial Neoplasia (CIN1).

DETAILED DESCRIPTION:
This study is to compare the regression rate of Cervical Intraepithelial Neoplasia (CIN1) between the treatment group and the control group.

The treatment group will be administered with PGA (Poly-gamma Glutamic Acid) for 4 weeks followed by 8 weeks observation.

The control group will be observed for 12 weeks without any comparator.

ELIGIBILITY:
Inclusion Criteria:

* Fertile women between age of 20 and 49
* Patients with cervical intraepithelial neoplasia 1(CIN1)
* HPV(Human Papilloma Virus) positive(+)
* White Blood Cell Count(WBC) over 4thous/ul, Hemoglobin above over 9.0g/dL Platelet over 150thous/uL and ANC(Absolute Neutrophil Count) over 1,500 10^6/L
* AST(Aspartate Aminotransferase) no less than 4 times higher than normal ALT(Alanine Aminotransferase) no less than 4 times higher than normal
* Normal for EKG(Electrocardiography) and no active disease detected trough chest X-ray
* Be informed of the nature of the study and will give written informed consent

Exclusion Criteria:

* Malignant tumor in any organ other than cervical intraepithelial neoplasia
* Active liver disease, immune disorder and severe renal failure
* Leukemia, collagenosis, sclerosis, autoimmune disease, clinically significant allergic disease(mild allergic symptom not required medicine excluded)
* Diagnosed diabetes
* Taking any of followings affecting immunological reaction within 7 days (Glucocorticoid, vitamins, health food and oriental medicine etc)
* Pregnancy and breastfeeding
* Registered in other clinical trials
* Patients whom the investigator considers inappropriate to participate in the study

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Regression rate | up to 12 weeks
  Regression rate will be assessed at the time of screening and 12 weeks. Regression means the change from the stage of CIN1 to normal.

SECONDARY OUTCOMES:
Reid Colposcopic Index | up to 12 weeks
  Reid Colposcopic Index will be assessed at the time of screening and 12 weeks.
Pap smear test | up to 12 weeks
  Result of Pap smear test will be assessed at the time of screening and 12 weeks.
HPV (Human Papilloma Virus) DNA Test | up to 12 weeks
  Result of HPV (Human Papilloma Virus) DNA Test will be assessed at the time of screening and 12 weeks.
HPV (Human Papilloma Virus) Hybrid CaptureII Test | up to 12 weeks
  Result of HPV (Human Papilloma Virus) Hybrid CaptureII Test will be assessed at the time of screening and 12 weeks.
NK (Natural Killer) Cell Activity | up to 12 weeks
  Result of NK (Natural Killer) Cell Activity will be assessed at the time of baseline (0day), 4 weeks, 8 weeks and 12 weeks.
Peripheral Blood Mononuclear Cells (PBMCs)Test | up to 12 weeks
  Result of Peripheral Blood Mononuclear Cells (PBMCs) Test will be assessed at the time of baseline (0day), 4 weeks, 8 weeks and 12 weeks.

OTHER OUTCOMES:
Adverse Events | up to 12 weeks
  Adverse events will be monitored for 12 weeks.
Vital Signs | up to 12 weeks
  Vital signs will be monitored for 12 weeks.
Laboratory Tests | up to 12 weeks
  Result of laboratory tests will be assessed at screening.

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Kwan Lee, MD, PhD, Principal Investigator — Korea University Guro Hospital; Tae Jin Kim, MD, PhD, Principal Investigator — Kwandong University College of Medicine Cheil Hospital; Jong Sup Park, MD, PhD, Principal Investigator — The Catholic University, Korea Seoul St Mary's Hospital; Chi-Heum Cho, MD, PhD, Principal Investigator — The Dongsan Medical Center of Keimyung University; Seok Ju Seong, MD, PhD, Principal Investigator — CHA University; Yongsoo Park, MD, PhD, Principal Investigator — MizMedi Hospital
Locations (7):
- South Korea (7):
  - Korea University Guro Hospital, Seoul, Seoul
  - The Dongsan Medical Center of Keimyung Hospital, Daegu
  - Kwandong University College of Medicine Cheil Hospital, Seoul
  - CHA Gangnam Hospital, Seoul
  - The Catholic University, Korea Seoul St Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - MiZMedi Hospital, Seoul

REFERENCES:
- [Derived] Cho HW, Park YC, Sung MH, Park JS, Kim TJ, Seong SJ, Cho CH, Lee JK. Short-term clinical and immunologic effects of poly-gamma-glutamic acid (gamma-PGA) in women with cervical intraepithelial neoplasia 1 (CIN 1): A multicenter, randomized, double blind, phase II trial. PLoS One. 2019 Jun 20;14(6):e0217745. doi: 10.1371/journal.pone.0217745. eCollection 2019. PMID 31220105